CLINICAL TRIAL: NCT03882294
Title: Effect of Probiotics and Its Associated Factors on Aflatoxin Biomarkers Among Healthy Subjects in Serdang and Kajang, Selangor: A Twelve-week Intervention
Brief Title: Probiotics and Its Associated Factors on Aflatoxin Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Rosita Jamaluddin, Associate Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO001
Record Dates: First submitted 2019-03-14; First posted 2019-03-20 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Aflatoxicosis
Keywords: probiotics; aflatoxin biomarkers; healthy subjects; intervention
MeSH Terms: conditions — Aflatoxin Poisoning | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized , double-blind, placebo-controlled, parallel trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care provider, and investigators will be blinded for the treatment assignment. A controller will be recruited to determine the two groups into probiotic and placebo groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Subjects in probiotic group will receive fermented milk containing live cultures Lactobacillus casei Shirota (LcS), 3 x 10^10 CFU/bottle (80 ml)
  Interventions: Other: Probiotics
- Placebo (Placebo Comparator): Subjects in placebo group will receive milk drink without LcS (80 ml).
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotics — Participants will be requested to consume the drinks (80 ml) twice a day - after lunch and dinner for 12 weeks.
  Arms: Probiotics
Other: Placebo — Participants will be requested to consume the drinks (80 ml) twice a day - after lunch and dinner for 12 weeks.
  Arms: Placebo

SUMMARY:
The study will be aimed to investigate the effect of probiotic intervention and its associated factors on aflatoxin biomarkers among healthy subjects in Serdang and Kajang, Selangor

DETAILED DESCRIPTION:
The study will be a randomized, double-blind, placebo-controlled, parallel intervention that conducted for 12 weeks and followed-up for 4 weeks among healthy adults under living condition in Serdang and Kajang, Selangor. 164 subjects will be recruited for the intervention study, where 82 subjects will be randomly allocated to the probiotic or placebo group. Probiotic and placebo drinks (80 ml) will be prepared in the form of bottle. Placebo drink will have similar taste, colour, physical appearance, and nutritional value as probiotic drink but contain no LcS. Morning urine samples (15 ml), weight status, and dietary intake will be collected every two weeks from week 0 to week 12 and follow up until week 16 at community centre. Whereas, fasting blood samples (5 ml) and physical activity will be collected every four weeks for 16 weeks at the community centre.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian healthy male or female adults (BMI <30kg/m2) aged 20 to 60 years who have regular bowel movement (at least 4 times/week), AFB1 >4.71 pg/mg albumin, and AFM1 > 0.88 ng/ml

Exclusion Criteria:

1. History or presence of any clinically important disease or disorder (eg. cardiovascular disease, kidney disease, diabetes mellitus, etc.) which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. Mental status that is incompatible with the proper conduct of the study
3. Functional constipation [based on Rome III diagnostic criteria with a five-point symptoms based diagnosing tool (0=never or rarely, 1=sometimes, 2=often, 3=most of the time, 4=always)]
4. Diarrhoea within 2 months prior to the study start
5. Allergic reaction towards probiotic, milk and with gastric problem
6. Lactose intolerance
7. Use of medications or/and antibiotics
8. Use of probiotic, prebiotic and fibre supplements or/and laxatives during the two weeks prior to study start.
9. Drug/alcohol abuse (for alcohol 4 times/day or 20 times/week)
10. Pregnant
11. Reported special diets such as vegetarian, vegan, or macrobiotic
12. Festive (eg. Ramadan, Chinese New Year etc) 3 months before and during the study
13. Participation in another intervention study one month prior to the present study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in serum AFB1-lysine adducts (pg/mg albumin) over 16 weeks | From week 0 to week 16
  Analysis of serum AFB1-lysine adducts will be done using elisa kit through HPLC.
Changes in urinary AFM1 (ng/ml) over 16 weeks | From week 0 to week 16
  Analysis of urinary AFM1 will be done using elisa kit.

SECONDARY OUTCOMES:
Changes in body mass index (kg/m^2) over 16 weeks | From week 0 to week 16
  Changes in weight and height will be measured using weighing scale and body meter respectively. Weight and height will be combined to report BMI in kg/m^2
Changes in waist circumference (cm) over 16 weeks | From week 0 to week 16
  The parameter will be measured using measuring tape.
Changes in physical activity level (MET-min/week) over 16 weeks | From week 0 to week 16
  The parameter will be examined using questionnaire based on the Global Physical Activity Questionnaire.
Changes in dietary intake over 16 weeks | From week 0 to week 16
  Dietary assessment will be recorded via food frequency questionnaire (FFQ). The conversion of food frequency to the amount of food intake is carried out using the following formula:
  Amount of food (g/day) = frequency of intake (conversion factor) × serving size × total of serving × weight of food in one serving (Wessex Institute of Public Health, 1995).
Changes in knowledge, attitude and practice (KAP) on aflatoxin over 16 weeks | From week 0 to week 16
  KAP will be examined using questionnaire in bilingual (English and Bahasa Malaysia). Knowledge towards aflatoxin is scored into two groups: know and do not know. Attitudes and practices are categorized using likert scale with 1=strongly disagree, 2=disagree, 3=agree and 4=strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Assoc Prof Dr Rosita Jamaluddin, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Teaching Hospital Universiti Putra Malaysia, Serdang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang WL, Akiyama T, Wang JS, Yong HY, Hassan F, Abu Saad H, Jamaluddin R, Sabran MR. Impact of Probiotic Lacticaseibacillus paracasei Strain Shirota (LcS) on Aflatoxin Exposure among Healthy Malaysian Adults: A Randomized, Double-Blind, Placebo-Controlled Intervention Study. J Nutr. 2025 Jul;155(7):2110-2121. doi: 10.1016/j.tjnut.2025.04.014. Epub 2025 Apr 16. PMID 40250564